CLINICAL TRIAL: NCT04180683
Title: Comparison Study of the Different Abbreviated Versions of the Geriatric Depression Scale (GDS) in Elderly With Neurocognitive Disorders Attending Social Responses
Brief Title: Comparison Study of the Different Abbreviated Versions of the Geriatric Depression Scale
Status: Completed | Type: Observational
Sponsor: Rsocialform - Geriatria, Lda (Other)
Responsible Party: Sponsor
Other Study IDs: 20112019
Record Dates: First submitted 2019-11-22; First posted 2019-11-27 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Depression; Depressive Disorder; Neurocognitive Disorders; Dementia
Keywords: Depression; Depressive Disorder; Neurocognitive Disorders; Dementia; Elderly; Geriatric Depression Scale; Beck Depression Inventory - II
MeSH Terms: conditions — Depression; Depressive Disorder; Neurocognitive Disorders; Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Semi-structured interview group: Participants assigned to this group will be administered the GDS-30, GDS-15, GDS-10 nad GDS-5, and also the BDI-II and a semi-structured interview based on the DSM-5 criteria. The psychologists performing the assessment will answer a questionnaire about which GDS version was more easily understandable by the participants and the participants' preference regarding the GDS versions.
  Interventions: Other: Battery of screening tests with semi-structured interview
- No semi-structured interview group: Participants assigned to this group will be administered the GDS-30 and the GDS-15, and also the BDI-II.
  Interventions: Other: Battery of screening tests without semi-structured interview

INTERVENTIONS:
Other: Battery of screening tests with semi-structured interview — First, participants will be administered the Mini-Mental State Examination to assess if they meet the inclusion criteria and an ID will be assigned to the participants that meet the criteria. Posteriorly, a clinical psychologist will administer the GDS-30, GDS-15, GDS-10 and GDS-5, the BDI-II and a semi-structured interview about depressive disorders according to the DSM-5 criteria. Participants with even ID's from each institution will be answer the instruments according to the order GDS-30, GDS-10, BDI-II, GDS-5 e GDS-15 and participants with odd ID's will answer the battery in the reverse order. The assessment session will take place in a single moment in time. After the assessment, the clinical psychologist will answer a questionnaire about which version was more easily understandable by the participants and the participants' preference regarding the GDS versions.
  Groups: Semi-structured interview group
Other: Battery of screening tests without semi-structured interview — First, participants will be administered the Mini-Mental State Examination to assess if they meet the inclusion criteria an ID will be assigned to the participants that meet the criteria. Posteriorly, a psychologist will administer the GDS-30, GDS-15 and the BDI-II. Participants with even ID's from each institution will answer the instruments according to the order GDS-30, BDI-II and GDS-15 and participants with odd ID's the administration order will answer the battery in the reverse order. The assessment session will take place in a single moment in time.
  Groups: No semi-structured interview group

SUMMARY:
This multicenter study conducted in several Portuguese institutions aims to compare the screening ability of the several Geriatric Depression Scale (GDS) validated versions for the Portuguese population (GDS-30, GDS-15, GDS-10 and GDS-5), as well as to establish their psychometric properties, using a large sample of elderly people with neurocognitive disorders attending social responses addressed to the elderly. Secondarily, cognitive state will be assessed.

DETAILED DESCRIPTION:
Depression is the most common mental health problem among older people, both in Portugal and around the world. Due to the fast aging of the world population, depression is a significant problem, with an estimated prevalence between 8% and 16%, which is more common in institutionalized elderly. Several studies have shown the negative consequences of depression in the elderly, which has been associated with higher morbidity and mortality rates, increased use of health services and increased costs. In addition, older people's depression is associated with major disability, chronic health problems, higher suicide rates, dementia and a lower quality of life. However, it is often an unrecognized, and therefore untreated, problem.

Under these circumstances, screening people at risk of depression (people with chronic illness, stroke, dementia, institutionalized or attending social responses, etc.) is a strategy with potential to reduce the impact of depression among the elderly.

One of the most commonly used screening scales for depressive symptoms in elderly is the Geriatric Depression Scale (GDS), a widely known and widely used scale designed specifically for older people. For this reason, it does not include questions related to somatic symptoms, as they lack discriminatory value in older people, because they can be attributed to other physical conditions or the aging process. The original version of the scale is composed by 30 items with a dichotomous response (yes/no) assessing motivation, energy, past and future orientation, mood, cognitive complaints, anxiety and irritability. The GDS scale has good psychometric properties and has been evaluated in a wide range of geriatric populations, institutionalized patients, elderly with chronic health problems, people with dementia, etc. In order to achieve better time efficiency in its administration, the original 30-item scale was abbreviated to a 15-item version. Posteriorly, multiple shorter versions of this scale were developed, composed by one, four, five, ten or twelve items.

The GDS scale has been widely translated and validated worldwide. In Portugal, the GDS-30 was adapted and validated by Pocinho, Farate, Dias, Lee and Yesavage. The versions of GDS-15, GDS-10 and GDS-5 were adapted and validated by Apóstolo and colleagues having demonstrated good psychometric properties and, therefore, potential as a screening tool for depressive symptoms in older people.

The aim of this study is to compare the screening ability of the several validated versions for the Portuguese population of the GDS scale (GDS-30, GDS-15, GDS-10 and GDS-5), as well as to establish their psychometric properties, using a large sample of elderly patients attending social responses addressed to the elderly. This study will allow recommendations on which is the most sensitive GDS version for detecting depressive symptoms by comparing them with other depression screening scales.

To achieve this, the results of the several GDS versions will be compared with the application of a gold standard, the Beck-II Depression Inventory [BDI-II].

Regarding the BDI-II, it is important to mention its good psychometric characteristics when used in the elderly population, which were evident in studies that compared the psychometric characteristics of different scales used to assess depression in the elderly. I was concluded that this instrument obtained a test-retest value of 0.93, Cronbach's α ranged from 0.76 to 0.91 in elderly Americans, in a community-dwelling elderly, in Puerto Rican residents, in elderly with heart problems, and in women living in institutions for the elderly. In elderly clinical samples, Cronbach's α ranged from 0.89 to 0.92. BDI is significantly and positively correlated with CES-D (r = 0.69, p <0.001) and with GDS (r = 0.71, p <0.001). The clinical utility of BDI-II is proven and high because of its clinical sensitivity and consistency with the DSM-IV criteria. In addition, it identifies many depressive symptoms and is one of the most commonly used instruments in the elderly without cognitive decline and also in non-clinical samples, as it is brief and easily administered and scored.

On the other hand, in another study where BDI-II was applied to elderly people with cognitive deficits, it was found that this population has symptoms similar to those of young people and adults, supporting the validity of this instrument in this population.

In order to reinforce the assessment of the screening ability of the several GDS versions validated for the Portuguese population, as well as to establish their psychometric properties, a sample (estimated at about 25%) will be defined, in which the GDS will be compared with a gold standard, that will consist of a semi-structured interview guide based on the criteria of the Diagnostic and Statistical Manual of Mental Disorders (5th ed.) for depressive disorders. For this sample, a questionnaire will be answered by the professionals who perform the evaluation, regarding their opinion about which GDS version is more easily understandable by the participants and the participants' preference regarding the different versions of GDS, as a means of assessing which version is more discernible for the participants. All the GDS versions validated for the Portuguese population (GDS-30, GDS-15, GDS-10 and GDS-5) will be administered to these participants.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of neurocognitive disorder according to the DSM-5 criteria and based on the MMSE scores.
* To be able to understand and answer the instruments' questions.
* Being 65 years of age or older.
* Being a native Portuguese speaker.
* To attend a social response addressed to the elderly in an institution.

Exclusion Criteria:

* Having severe sensory and physical limitations, severe disconnection from the environment, or presence of severe neuropsychiatric symptoms that make it impossible to administer the assessment battery.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: In each participanting institution, users who meet the inclusion criteria will be selected to answer the assessment instruments. Prior to the inclusion in the study, informed consent will be obtained from participants or their caregivers after they have received information about the study. This information will include the purpose of the study, the data processing in accordance with current legislation, the voluntary nature of the participation in the study and the right to withdraw consent at any time without affecting the services received in the institution.
Sampling Method: Non-Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Depressive symptomatology assessed through the GDS-30 | Baseline
  Participants' scores in the GDS-30. This instrument evaluated depressive symptoms using yes/no answers. Scores range between 0 and 30 points. Higher scores indicate more severe depressive symptoms.
Depressive symptomatology assessed through the GDS-15 | Baseline
  Participants' scores in the GDS-15. This instrument evaluated depressive symptoms using yes/no answers. Scores range between 0 and 15 points. Higher scores indicate more severe depressive symptoms.
Depressive symptomatology assessed through the GDS-10 | Baseline
  Participants' scores in the GDS-10. This instrument evaluated depressive symptoms using yes/no answers. Scores range between 0 and 10 points. Higher scores indicate more severe depressive symptoms.
Depressive symptomatology assessed through the GDS-5 | Baseline
  Participants' scores in the GDS-5. This instrument evaluated depressive symptoms using yes/no answers. Scores range between 0 and 5 points. Higher scores indicate more severe depressive symptoms.
Depressive symptomatology assessed through the BDI-II | Baseline
  Participants' scores in the BDI-II. This instrument evaluates depressive symptoms. Scores range from 0 to 63 points. Higher scores indicate more severe depressive symptoms.
Depressive symptomatology assessed through the semi-structured interview | Baseline
  Participants' answers in the semi-structured interview. This interview includes questions regarding depressive symptomatology and is based on the DSM-5 criteria.

SECONDARY OUTCOMES:
Cognitive state evaluated through the Mini-Mental State Examination | Baseline
  Participants' scores/answers in the MMSE that will allow to understand if the participants meet the inclusion criteria. MMSE is a brief cognitive screening test. Scores range between 0 - 30 points. Higher scores indicate better cognitive function. MMSE will be administered to all participants.
Acceptability of the instruments by the participants evaluated though the questionnaire applied to the psychologists | Baseline
  Psychologists answers in the questionnaire, designed specifically for this study. It will allow to understand which version is more easily understandable by the participants and their preference regarding the GDS versions. This questionnaire will only be answered by the clinical psychologists that conducted the evaluation sessions with the participants in the Semi-structured interview group.

OTHER OUTCOMES:
Sociodemographic information gathered through the sociodemographic questionnaire | Baseline
  Participants' answers in the sociodemographic questionnaire designed specifically for this study. It gathers information about gender, age, marital status, formal education, which social response the participant attends, medical comorbidities and cognitive symptoms and will be administered to all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Susana I Justo Henriques, PhD, Principal Investigator — Cediara and Nursing School of Coimbra; Enrique Pérez Saéz, PhD, Principal Investigator — CRE Alzheimer and University of Salamanca; João L Alves Apóstolo, PhD, Principal Investigator — Nursing School of Coimbra; Patrícia Otero Otero, PhD, Principal Investigator — Universidade da Coruña; Fernando L Vázquez González, PhD, Principal Investigator — University of Santiago de Compostela
Locations (32):
- Portugal (32):
  - Cediara - Associação de Solidariedade Social de Ribeira de Fráguas, Albergaria-a-Velha, Aveiro District
  - Rsocialform - Geriatria, Lda., Mealhada, Aveiro District
  - Centro de Assistência Paroquial da Pampilhosa, Mealhada, Aveiro District
  - Fundação Luiz Bernardo de Almeida, Vale de Cambra, Aveiro District
  - Lar D. Pedro V, Praia da Vitória, Azores
  - Santa Casa da Misericórdia de Ferreira do Alentejo, Ferreira do Alentejo, Beja District
  - Centro Social e Paroquial de S. Martinho de Medelo, Fafe, Braga District
  - Centro Social Vale do Homem, Vila Verde, Braga District
  - Lar de S. José, Covilha, Castelo Branco District
  - Santa Casa da Misericórdia do Fundão, Fundão, Castelo Branco District
  - PRODECO - Progresso e Desenvolvimento de Covões, Cantanhede, Coimbra District
  - Fundação Sarah Beirão/António Costa Carvalho, Tábua, Coimbra District
  - Santa Casa da Misericórdia de Alcobaça, Alcobaça, Leiria District
  - Santa Casa da Misericórdia de Alvorge, Ansião, Leiria District
  - Centro Social e Paroquial de S. Vicente de Alcabideche, Alcabideche, Lisbon District
  - Fundação AFID Diferença, Amadora, Lisbon District
  - Irmãs Hospitaleiras - Casa de Saúde da Idanha, Sintra, Lisbon District
  - Santa Casa da Misericórdia de Arronches, Arronches, Portalegre District
  - Santa Casa da Misericórdia de Arez, Nisa, Portalegre District
  - Associação de Solidariedade Social de Ponte de Sôr, Ponte de Sôr, Portalegre District
  - Quintinha da Conceição Sousa & Silva Lda, Maia, Porto District
  - Centro Social Paroquial de Recarei, Paredes, Porto District
  - Associação de Desenvolvimento da Vila de Paço Sousa, Penafiel, Porto District
  - Centro Social de Bem-Estar de Alcanena, Alcanena, Santarém District
  - Santa Casa da Misericórdia de Canha, Montijo, Setúbal District
  - Santa Casa da Misericórdia de Caminha, Caminha, Viana do Castelo District
  - Santa Casa da Misericórdia de Melgaço, Melgaço, Viana do Castelo District
  - Santa Casa da Misericórdia de Tarouca, Tarouca, Viseu District
  - Santa Casa da Misericórdia de Vouzela, Vouzela, Viseu District
  - Santa Casa da Misericórdia de Castelo Branco, Castelo Branco
  - Cáritas de Coimbra, Coimbra
  - Fundação João Bento Raimundo, Guarda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson DN. Treating depression in old age: the reasons to be positive. Age Ageing. 2001 Jan;30(1):13-7. doi: 10.1093/ageing/30.1.13. PMID 11322666
- [Background] ApóstoloJ, Bobrowicz-Campos E, Reis I, Henriques S, Correia C. Screening capacity of Geriatric Depression Scale with 10 and 5 items. Revista de Enfermagem Referência, 4(16): 29-38, 2018. doi:10.12707/RIV17062
- [Background] Apóstolo JLA, Bobrowicz-Campos EM, Reis IA, Henriques SJ, Correia CAV. Exploring the screening capacity of the European Portuguese version of the 15-item Geriatric Depression Scale. Revista de Psicopatología y Psicología Clínica, 23(2): 99, 2018. doi:10.5944/rppc.vol.23.num.2.2018.21050
- [Background] Apóstolo J, Loureiro L, Reis I, Silva I, Cardoso D, Sfetcu R. Contribution to the adaptation of the Geriatric Depression Scale -15 into Portuguese. Revista de Enfermagem Referência, IV(3): 65-73, 2014. doi:10.12707/RIV14033
- [Background] Balsamo M, Cataldi F, Carlucci L, Padulo C, Fairfield B. Assessment of late-life depression via self-report measures: a review. Clin Interv Aging. 2018 Oct 16;13:2021-2044. doi: 10.2147/CIA.S178943. eCollection 2018. PMID 30410319
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] Birrer RB, Vemuri SP. Depression in later life: a diagnostic and therapeutic challenge. Am Fam Physician. 2004 May 15;69(10):2375-82. PMID 15168957
- [Background] Blazer DG. Depression in late life: review and commentary. J Gerontol A Biol Sci Med Sci. 2003 Mar;58(3):249-65. doi: 10.1093/gerona/58.3.m249. PMID 12634292
- [Background] Campos RC, Gonçalves B. The Portuguese version of the Beck Depression Inventory-II (BDI-II): Preliminary psychometric data with two nonclinical samples. European Journal of Psychological Assessment, 27(4): 258-264, 2011. doi:10.1027/1015-5759/a000072
- [Background] Carvalho JO, Tan JE, Springate BA, Davis JD. Self-reported depressive syndromes in mild cognitive impairment and mild Alzheimer's disease. Int Psychogeriatr. 2013 Mar;25(3):439-44. doi: 10.1017/S1041610212001676. Epub 2012 Oct 19. PMID 23083490
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Freitas S, Simoes MR, Alves L, Santana I. The Relevance of Sociodemographic and Health Variables on MMSE Normative Data. Appl Neuropsychol Adult. 2015;22(4):311-9. doi: 10.1080/23279095.2014.926455. Epub 2014 Dec 22. PMID 25531579
- [Background] Guerreiro M, Silva AP, Botelho MA, Leitão O, Castro-Caldas A, Garcia C. Adaptação à população portuguesa da tradução do Mini Mental State Examination (MMSE). Revista Portuguesa de Neurologia, 1(9): 9-10, 1994.
- [Background] Jongenelis K, Pot AM, Eisses AM, Gerritsen DL, Derksen M, Beekman AT, Kluiter H, Ribbe MW. Diagnostic accuracy of the original 30-item and shortened versions of the Geriatric Depression Scale in nursing home patients. Int J Geriatr Psychiatry. 2005 Nov;20(11):1067-74. doi: 10.1002/gps.1398. PMID 16250079
- [Background] Morgado J, Rocha C, Maruta C, Guerreiro M, Martins I. Novos valores normativos do mini-mental state examination. Sinapse, 9, (2): 10-16, 2009.
- [Background] Pocinho MTS, Farate C, Dias CA, Lee TT, Yesavage JA. Clinical and Psychometric Validation of the Geriatric Depression Scale (GDS) for Portuguese Elders. Clinical Gerontologist, 32(2): 223-236, 2009. doi:10.1080/07317110802678680
- [Background] Pocklington C, Gilbody S, Manea L, McMillan D. The diagnostic accuracy of brief versions of the Geriatric Depression Scale: a systematic review and meta-analysis. Int J Geriatr Psychiatry. 2016 Aug;31(8):837-57. doi: 10.1002/gps.4407. Epub 2016 Feb 18. PMID 26890937
- [Background] Sheikh JL, Yesavage JA. Geriatric depression scale (GDS): Recent evidence and development of a shorter version. In T. L. Brink (Ed.), Clinical gerontology: A guide to assessment and intervention. New York: Hawthorne Press, 1986.
- [Background] de Sousa RD, Rodrigues AM, Gregorio MJ, Branco JDC, Gouveia MJ, Canhao H, Dias SS. Anxiety and Depression in the Portuguese Older Adults: Prevalence and Associated Factors. Front Med (Lausanne). 2017 Nov 20;4:196. doi: 10.3389/fmed.2017.00196. eCollection 2017. PMID 29209612
- [Background] Weeks SK, McGann PE, Michaels TK, Penninx BW. Comparing various short-form Geriatric Depression Scales leads to the GDS-5/15. J Nurs Scholarsh. 2003;35(2):133-7. doi: 10.1111/j.1547-5069.2003.00133.x. PMID 12854293
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Zhao K, Bai ZG, Bo A, Chi I. A systematic review and meta-analysis of music therapy for the older adults with depression. Int J Geriatr Psychiatry. 2016 Nov;31(11):1188-1198. doi: 10.1002/gps.4494. Epub 2016 Apr 19. PMID 27094452